CLINICAL TRIAL: NCT04175054
Title: Training to Restore Walking and Promote Nervous System Repair in Multiple Sclerosis: RCT to Determine the Importance of Intensity
Brief Title: Comparison of Vigorous Versus Low Intensity Cool Room Treadmill Training in People with Multiple Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study no longer feasible.
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Michelle Ploughman, Associate Professor of Medicine, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20201156
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Neurological Rehabilitation; Exercise; Neuronal Plasticity; Cooling
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is an assessor-blinded Randomized Controlled Trial.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to group allocation, and will not be involved in conducting the training intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Intensity Group (Active Comparator): Less than 40% Heart Rate Reserve
  Interventions: Other: Body-weight supported treadmill training in a room cooled to 16°C
- Vigorous Intensity Group (Experimental): More than 60% Heart Rate Reserve
  Interventions: Other: Body-weight supported treadmill training in a room cooled to 16°C

INTERVENTIONS:
Other: Body-weight supported treadmill training in a room cooled to 16°C — Exercise will be performed on a treadmill using an overhead harness for safety in a temperature controlled-room at 16°C with 1:1 supervision. The high intensity group will maintain vigorous intensity with a target workload >60% of heart rate reserve for 30 min (plus 5min warm up and 5min cool down) while the low-intensity group will walk at mild intensity (<40% heart rate reserve) for the same duration. Heart rate, blood pressure, and rating of perceived exertion will be recorded throughout to monitor for potential adverse events and to ensure that target training zone heart rates are maintained. The intervention is 3 times per week for 12 weeks, with a 3-month run-in observational period to confirm disease stability, and 3-month follow-up to determine the sustainability of effects.

SUMMARY:
New research in animal models of MS suggests that greater training intensity is required to restore lost functions. We have developed and tested vigorous intensity cool room treadmill training that people with MS who have fatigue and heat-sensitivity can tolerate. This study will focus on the appropriate dosage of training.

DETAILED DESCRIPTION:
Our previous research showed that vigorous aerobic training in a room cooled to 16°C can improve walking and measures of brain plasticity among people with MS related walking disability, especially in those who had fatigue and heat sensitivity. As a next step, we will compare our novel vigorous intensity cool room treadmill training to low intensity cool room treadmill walking and determine whether intensity is important in order to improve brain repair and restore walking among people with MS. Our first objective is to compare the effects of 12 weeks of vigorous versus low intensity training on walking. Our second objective is to determine whether treadmill training alters indicators of brain repair. We hypothesize that the cool room vigorous training will result in greater increases in walking and less fatigue, which will be sustained at follow-up. We also hypothesize that improvements will align with less brain inhibition (shortened CSP measured using Transcranial Magnetic Stimulation) and greater upregulation of the neurotrophin IGF-1.

ELIGIBILITY:
Inclusion Criteria:

* people with a confirmed diagnosis of relapsing-remitting or progressive MS
* older than 18 and less than 70 years of age
* able to walk at least 10 meters with use of walking aids (Expanded Disability Status Scale (EDSS) <7.0)
* must be stable without relapse for at least 90 days

Exclusion Criteria:

* currently attending physical rehabilitation
* functional community ambulators (gait speed>120 cm/s)
* a relapse of MS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2030-01 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Fast walking speed | 12 weeks
  Gait velocity (cm/s) measured while walking at fast pace

SECONDARY OUTCOMES:
Spatiotemporal parameters of gait measured while walking at self-selected pace | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  Walkway outputs include step length and width (cm), double support time (%), symmetry (ratio between affected and less-affected sides)
Maximal oxygen consumption during graded exercise test | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  VO2max
Multiple Sclerosis Impact Scale-29 | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  The Multiple Sclerosis Impact Scale-29 provides physical and psychological sub-scales. Using a Likert scale, participants indicate the degree to which problems, such as 'moving about' and 'balance' affect them from 'not at all' to 'extremely'.
Fatigue Severity Scale | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  A 9-item questionnaire, which assesses the severity of fatigue with items scored on a 7-point scale, '1 = strongly disagree' and '7 = strongly agree'. The minimum and maximum score possible are 9 and 63 respectively. Another reporting method is the mean of all scores from all 9-items, with minimum and maximum score possible being 1 and 7 respectively.
Hospital Anxiety and Depression Scale | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  A self-reported rating scale of severity of mood symptoms ranging from 0-21 with higher score indicating more symptoms.
Montreal Cognitive Assessment | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  Measures overall cognitive function with score ranging from 0 to 30 with higher scores indicating higher executive function
Symbol Digit Modality Test | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  Cognitive impairment
Transcranial Magnetic Stimulation | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  Corticospinal excitability
Serum Insulin-like growth factor-1 (IGF-1) | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  Resting and exercise-induced serum levels of IGF-1 in response to the 12-week exercise intervention
Structural and functional brain changes on Magnetic Resonance Imaging (MRI) | Following completion of the 12-week exercise intervention and 3-months post-exercise intervention
  Standardized protocol recommended by the Canadian Dementia Imaging Group (https://www.cdip-pcid.ca/) which includes T1 and T2-weighted structural images, diffusion tensor imaging, and resting state connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ploughman, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No